CLINICAL TRIAL: NCT02501135
Title: A Retrospective Investigation of Safety and Efficacy From Increasing Concentrations of Local Anesthetic in Pediatric Femoral Nerve Blocks
Brief Title: A Retrospective Investigation of Local Anesthetic Concentrations in Femoral Nerve Block
Status: Completed | Type: Observational
Sponsor: Giorgio Veneziano (Other)
Responsible Party: Sponsor-Investigator, Giorgio Veneziano, Clinical Assistant Professor, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: IRB 15-00396
Record Dates: First submitted 2015-05-28; First posted 2015-07-17 (Estimated); Results first posted 2019-03-06 (Actual); Last update posted 2019-03-06 (Actual); Status verified 2018-11

CONDITIONS: Postoperative Pain
Keywords: Femoral nerve blocks; children; knee and thigh surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Ropivacaine; Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Femoral Nerve Blocks: Patients who receive ropivacaine or bupivacaine during femoral nerve block.
  Interventions: Procedure: Femoral nerve block with ropivacaine or bupivacaine

INTERVENTIONS:
Procedure: Femoral nerve block with ropivacaine or bupivacaine

SUMMARY:
The purpose of this study is to retrospectively compare perioperative pain relief and safety in pediatric patients who have received a femoral nerve block with varying concentrations of local anesthetic.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II
* Age < or equal to 18 years of age at time of femoral nerve block
* Femoral nerve block performed from 2010-2015

Exclusion Criteria:

* ASA physical status > II
* Co-morbid diseases (cardiac, pulmonary, neurological disease)
* Use of adjunctive medications in femoral nerve block (except for epinephrine), such as dexamethasone

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who have undergone anesthesia and received a femoral nerve block at Nationwide Children'ts Hospital from 2010-2015 utilizing our EMR - PICIS.
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2015-06; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giorgio Veneziano, MD, Principal Investigator — Nationwide Children's Hospital

RESULTS

PARTICIPANT FLOW:
Groups:
- Femoral Nerve Blocks: Patients who receive ropivacaine or bupivacaine during femoral nerve block.
  Femoral nerve block with ropivacaine or bupivacaine
Period: Overall Study
Arm/Group | Femoral Nerve Blocks
Started | 281
Completed | 281
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Femoral Nerve Blocks
Number analyzed (Participants) | 281
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 281
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 14.5 [13 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 172
Region of Enrollment [Number; unit: participants]
  United States | 281

OUTCOME MEASURES:

1. Primary Outcome: Concentration of Local Anesthetic Injected for Femoral Nerve Block
Time Frame: length of surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Femoral Nerve Blocks
Number analyzed (Participants) | 281
Participants
  Patients who received ropivacaine 0.2% | 117
  Patients who received ropivacaine 0.5% | 81
  Patients who received bupivacaine 0.25% | 83

2. Primary Outcome: Total mg of Local Anesthetic Injected for Femoral Nerve Block
Time Frame: length of surgery
Measure: Median (Inter-Quartile Range); unit: ml/kg
Groups:
- Femoral Nerve Blocks: Patients who receive ropivacaine or bupivacaine during femoral nerve block.
  Amount of femoral nerve block with ropivacaine or bupivacaine
Arm/Group | Femoral Nerve Blocks
Number analyzed (Participants) | 281
ml/kg
  Amount of ropivacaine 0.2% | 0.27 [0.22 to 0.35]
  Amount of ropivacaine 0.5% | 0.29 [0.22 to 0.35]
  Amount of bupivacaine 0.25% | 0.25 [0.19 to 0.32]

3. Primary Outcome: Intraoperative Tylenol Administered
Description: Amount of Tylenol administered based on if got ropivacaine or bupivacaine femeral nerve block.
Time Frame: length of surgery
Measure: Number; unit: percentage of participants
Groups:
- Intraoperative Tylenol Consumption: Patients who receive ropivacaine or bupivacaine during femoral nerve block and their Tylenol consumptiong during surgery
Arm/Group | Intraoperative Tylenol Consumption
Number analyzed (Participants) | 281
percentage of participants
  Increased Tylenol use in ropivacaine 0.5% NB | 16
  Increased Tylenol use in ropivacaine 0.2% NB | 4
  Increased Tylenol use in bupivacaine 0.25% NB | 1

4. Primary Outcome: Post-operative Opioids Administered
Description: Amount of opioid consumption in the post operative anesthesia care unit depending on if the patient received femoral nerve block with ropivacaine or bupivacaine
Time Frame: in PACU (1 hr post-op)
Measure: Median (Inter-Quartile Range); unit: mg/kg
Groups:
- Post Operative Opioid Consumption: Patients who receive ropivacaine or bupivacaine during femoral nerve block and their opioid consumption in PACU
Arm/Group | Post Operative Opioid Consumption
Number analyzed (Participants) | 281
mg/kg
  IV Morphine who got ropivacaine 0.5% nerve block | 0 [0 to 0.04]
  IV Morphine who got ropivacaine 0.2% nerve block | 0.02 [0 to 0.07]
  IV Morphine who got bupivacaine 0.25% nerve block | 0.02 [0 to 0.08]

5. Secondary Outcome: Time to Discharge From PACU
Time Frame: Conclusion of surgery until admission to assigned unit or to phase, an expected average of 1 hour
Population: One patient was excluded from analysis of time to PACU discharge due to a missing PACU arrival time.
Measure: Median (Inter-Quartile Range); unit: minutes
Groups:
- Discharge From PACU in Minutes: The amount of time spent in the post-anesthesia care unit (PACU) in minutes
Arm/Group | Discharge From PACU in Minutes
Number analyzed (Participants) | 280
minutes
  PACU time in pt who got ropivacaine 0.2% | 57 [41 to 76]
  PACU time in pt who got ropivacaine 0.5% | 47 [36 to 68]
  PACU time in pt who got bupivacaine 0.25% | 55 [35 to 80]

6. Secondary Outcome: Post-operative Pain Scale Using FLACC
Description: The Face, Legs, Activity, Cry, Consolability scale or FLACC scale is a measurement used to assess pain for children between the ages of 2 months and 7 years or individuals that are unable to communicate their pain. The scale is scored in a range of 0-10 with 0 representing no pain.
Time Frame: 1 hour post-op
Population: 63 of the 281 total subjects had their pain assessed using the FLACC pain scale.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- FLACC Pain Scores: Patients who receive ropivacaine or bupivacaine during femoral nerve block and their FLACC pain scores
Arm/Group | FLACC Pain Scores
Number analyzed (Participants) | 63
units on a scale
  FLACC in patient who had ropivacaine 0.2% | 0 [0 to 2]
  FLACC in patient who had ropivacaine 0.5% | 0 [0 to 0]
  FLACC in patient who had bupivacaine 0.25% | 0 [0 to 0]

7. Secondary Outcome: Post-operative Pain Scale Using VAS
Description: The visual analogue scale (VAS) for pain is a validated, subjective measure where scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Time Frame: 1 hour post-op
Population: 197 out of the total 281 subjects had their pain assessed using VAS.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Groups:
- VAS Pain Scores: Patients who receive ropivacaine or bupivacaine during femoral nerve block and their VAS pain scores
Arm/Group | VAS Pain Scores
Number analyzed (Participants) | 197
units on a scale
  Ropivacaine 0.2% | 0 [0 to 5]
  Ropivacaine 0.5% | 0 [0 to 4]
  Bupivacaine 0.25% | 0 [0 to 6]

ADVERSE EVENTS:
Arm/Group | Femoral Nerve Blocks
All-Cause Mortality (participants affected / at risk) | 0/281
Serious Adverse Events (participants affected / at risk) | 0/281
Other Adverse Events (participants affected / at risk) | 0/281

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2015-05-21): https://cdn.clinicaltrials.gov/large-docs/35/NCT02501135/Prot_000.pdf